CLINICAL TRIAL: NCT03755232
Title: Determination of the Acute Glycemic and Insulinemic Response of FOSSENCE™ Alone, or When Substituted or Added to a Carbohydrate Challenge: A Three-phase, Acute, Randomized, Cross-over, Double Blind Clinical Trial
Brief Title: Acute Glycemic and Insulinemic Response of FOSSENCE™
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TATA CHEMICALS LTD (Industry)
Collaborators: Glycemic Index Laboratories, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GIL-1841Tata
Record Dates: First submitted 2018-11-23; First posted 2018-11-27 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Dietary Modification; Healthy
Keywords: dietary fibre; fructo-oligosaccharide; prebiotic; glucose metabolism; insulin metabolism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- scFOS treatment #1 (Experimental): Phase 1: 10g of scFOS Phase 2: 50g dextrose +15g scFOS Phase 3: 50g avCHO from white bread +15g scFOS
  Interventions: Dietary Supplement: scFOS
- scFOS treatment #2 (Experimental): Phase 1: n/a Phase 2: 35g Dextrose +15g scFOS Phase 3: 35g avCHO from white bread +15g scFOS
  Interventions: Dietary Supplement: scFOS
- Control #1 (Active Comparator): Phase 1: Water control (negative control) Phase 2: 35g Dextrose control 1 Phase 3: 35g avCHO from white bread (control 1)
  Interventions: Other: Control
- Control #2 (Active Comparator): Phase 1: 10g Dextrose (positive control) Phase 2: 50g Dextrose control 2 Phase 3: 50g avCHO from white bread (control 2)
  Interventions: Other: Control

INTERVENTIONS:
Dietary Supplement: scFOS — Fossence™ (short chain Fructo-oligosaccharides (scFOS)
  Arms: scFOS treatment #1; scFOS treatment #2
Other: Control — water or dextrose or white bread
  Arms: Control #1; Control #2

SUMMARY:
Short chain fructooligosaccharide (FOS) is known as a prebiotic fiber/nutrient and has been documented to demonstrate different health benefits including glucose control, gut health, mineral absorption, weight and immunity.

FossenceTM is a short chain fructo-oligosaccharide (scFOS), sweet tasting, soluble prebiotic dietary fibre which is produced through Tata Chemicals Limited's patented process and is currently US GRAS notified (safe for consumption). The formulation and properties of scFOS suggest that the molecule may potentially play a role in glucose and insulin metabolism.

The purpose of this study is to explore the rise of glucose and insulin in the blood after consuming FossenceTM that has been added or substituted into a sugar drink or white bread.

DETAILED DESCRIPTION:
BACKGROUND Short chain fructooligosaccharide (FOS) is known as a prebiotic fiber/nutrient and has been documented to demonstrate different health benefits including attenuation of postprandial glycemia, gut health, mineral absorption, satiety & weight management and immunity.

FossenceTM is short chain fructo-oligosaccharide (scFOS), a sweet tasting, soluble dietary fibre which is produced through Tata Chemicals Limited's patented process. These properties of scFOS suggest that the molecule may potentially play a role in glucose and insulin metabolism. The proposed 3 phase study will therefore explore the properties of FossenceTM with respect to its fibre like properties (not digested in the human small intestine), and its effect on postprandial glycemia when added or substituted into a simple (dextrose) or complex (white bread) carbohydrate load.

OBJECTIVES The purpose of this 3 phase study is to: 1. Demonstrate that consumption of scFOS does not increase postprandial blood glucose levels, 2. Explore the effects when scFOS is either added or substituted into a simple carbohydrate load (dextrose) or 3. Into a complex carbohydrate food (white bread).

PARTICIPANTS Twenty five healthy adult males and non-pregnant, non-lactating females, aged 18-65 years with BMI between 18 and 30 kg/m2 are required for each phase.

DESIGN The study is a double-blind, randomized, cross-over trial.

POWER CALCULATION Using the t-distribution and assuming an average coefficient of variation (CV) of within-individual variation of 2-hour glucose incremental are under the curve (IAUC) values of 23%, n=25 subjects has 90% power to detect a 22% difference in 2-hour glucose IAUC with 2-tailed p<0.05.

Using the t-distribution and assuming an average CV of within-individual variation of 2-hour insulin IAUC values of 25%, n=25 subjects has 90% power to detect a 24% difference in 2-hour insulin IAUC with 2-tailed p<0.05.

RECRUITMENT Participants will be recruited from the pool of participants at Glycemic Index Laboratories (GI Labs) who have indicated that they are willing to be contacted and asked if they wish to participate in new studies. If an insufficient number of subjects can be recruited, then an advertisement will be used to recruit new subjects.

INTERVENTIONS

Phase 1: to assess the glucose and insulin responses to the following test meals:

1. 10g of scFOS
2. A negative control (water)
3. A positive control (10g of dextrose)

Phase 2: to assess the glucose and insulin responses to the following test meals:

1. 50g Dextrose +15g scFOS,
2. 35g Dextrose +15g scFOS,
3. 35g Dextrose and
4. 50g Dextrose.

Phase 3: to assess the glucose and insulin responses to the following test meals:

1. 50g available carbohydrate (avCHO) from white bread +15g scFOS,
2. 35g avCHO from white bread +15g scFOS,
3. 35g avCHO from white bread and
4. 50g of avCHO from white bread

STATISTICAL ANALYSIS

For each study phase the following will be the statistical method:

Data will be presented as mean, standard deviation (SD) and standard error of the mean (SEM) values.

The mean glucose or insulin concentration in the 2 fasting blood samples will be used as the fasting concentration for the purposes of calculating incremental areas under the glucose and serum insulin response curves (IAUC), ignoring area below fasting17. Glucose and insulin concentrations, glucose and insulin IAUC (from 0 to 120 minutes) will be subjected to repeated measures analysis using the General Linear Model of variance (GLM-ANOVA). After demonstration of significant heterogeneity, the significance of differences among individual means will be determined using Tukey's method with p<0.05. In addition, differences at individual time points for glucose and insulin will be assessed. Differences will be considered to be statistically significant if 2-tailed p<0.05.

OUTCOMES

The primary analysis of each phase will be:

Phase 1: to compare the incremental area under the glucose curve elicited by

1. 10g of scFOS
2. A negative control (water)
3. A positive control (10g of dextrose)

Phase 2: to compare the incremental areas under the glucose curve elicited by

1. 50g Dextrose +15g scFOS,
2. 35g Dextrose +15g scFOS,
3. 35g Dextrose and
4. 50g Dextrose.

Phase 3: to compare the incremental areas under the glucose curve elicited by

1. 50g available carbohydrate (avCHO) from white bread +15g scFOS,
2. 35g avCHO from white bread +15g scFOS,
3. 35g avCHO from white bread and
4. 50g of avCHO from white bread

The secondary analyses of each phase will be:

Phase 1: to compare the glucose and insulin levels at individual time points, and the incremental area under the serum insulin curve elicited by 10g of scFOS with a negative control (water) or positive control (10g of dextrose)

Phase 2: to compare the glucose and insulin levels at individual time points, and the incremental area under the serum insulin curve elicited by:

(4) 50g Dextrose +15g scFOS, (5) 35g Dextrose +15g scFOS, (6) 35g Dextrose and (7) 50g Dextrose.

Phase 3: to compare the glucose and insulin levels at individual time points and the incremental area under the serum insulin curve elicited by:

1. 50g available carbohydrate (avCHO) from white bread +15g scFOS,
2. 35g avCHO from white bread +15g scFOS,
3. 35g avCHO from white bread and
4. 50g of avCHO from white bread

ELIGIBILITY:
Subjects (N= 25) will be men (at least N= 12) and non-pregnant, non-lactating women (at least N= 12), 18 - 65 years of age each with a BMI of 18 - 30 kg/m2 inclusive and

Inclusion Criteria:

* Blood pressure < 140/90 mmHg
* No major illness or surgery requiring hospitalization within 3 months of the first study visit after screening
* No history of cardiovascular, metabolic, respiratory, renal, gastrointestinal or hepatic disease
* Subject may be a male or a non-pregnant, non-lactating female, at least 6 weeks postpartum prior to screening visit
* Willing to maintain habitual diet, physical activity pattern, and body weight throughout the study
* Subjects must be eligible to receive income in Canada and must demonstrate Ontario Health Insurance Program coverage

Exclusion Criteria:

* Failure to meet all the inclusion criteria
* Previous bariatric procedure
* No chronic disease such as type-1 or type-2 diabetes mellitus (fasting blood sugar levels <100 mg/dL (or <5.6 mmol/L) as assessed at the first visit)
* No gastro-intestinal disorder such as Crohn's disease, coeliac disease, irritable bowel syndrome
* Medications known to affect glucose tolerance -but stable doses of oral contraceptives, acetylsalicylic acid, thyroxin, vitamins and mineral supplements or drugs to treat hypertension, hyperlipidemia, anxiety/depression or osteoporosis are acceptable
* Any known food allergies or intolerances
* No strong dislike of or intolerance to sweetened beverages or inulin
* Smokers
* Alcohol consumption of no more than 10 drinks per week for women and 15 drinks per week for men. One drink is defined as either 5oz wine, 341ml of beer/cider or 1.5 oz distilled alcohol
* History of cancer in the prior two years, except for non-melanoma skin cancer
* Participants who do not understand English
* Presence of any condition, illness or drug use, which in the opinion of Dr. Wolever, increases the risk to the subject or to others or may affect the results

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2019-02-27 (Actual); Study Completion 2019-09-09 (Actual)

PRIMARY OUTCOMES:
incremental area under the 2 hour (120 minutes) blood glucose curve | 0-120 minutes
  The mean glucose concentration in the 2 fasting blood samples will be used as the fasting concentration for the purposes of calculating incremental area under the glucose response curve (IAUC), ignoring area below fasting

SECONDARY OUTCOMES:
incremental area under the 2 hour (120 minutes) blood insulin curve | 0-120 minutes
  The mean insulin concentration in the 2 fasting blood samples will be used as the fasting concentration for the purposes of calculating incremental area under the insulin response curve (IAUC), ignoring area below fasting
comparison of the glucose and insulin levels at individual time points from 0-120min | 0-120 minutes
  to compare the glucose and insulin levels at individual time points (at -fasting, 15, 30, 45, 60, 90 and 120 min (7 time points)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas MS Wolever, MD, Principal Investigator — Glycemic Index Laboratories, Inc
Locations (1):
- INQUIS Clinical Research (formerly GI Labs), Toronto, Ontario, Canada

REFERENCES:
- [Background] Bouhnik Y, Raskine L, Simoneau G, Paineau D, Bornet F. The capacity of short-chain fructo-oligosaccharides to stimulate faecal bifidobacteria: a dose-response relationship study in healthy humans. Nutr J. 2006 Mar 28;5:8. doi: 10.1186/1475-2891-5-8. PMID 16569219
- [Background] Bouhnik Y, Raskine L, Simoneau G, Vicaut E, Neut C, Flourie B, Brouns F, Bornet FR. The capacity of nondigestible carbohydrates to stimulate fecal bifidobacteria in healthy humans: a double-blind, randomized, placebo-controlled, parallel-group, dose-response relation study. Am J Clin Nutr. 2004 Dec;80(6):1658-64. doi: 10.1093/ajcn/80.6.1658. PMID 15585783
- [Background] Du H, van der A DL, Boshuizen HC, Forouhi NG, Wareham NJ, Halkjaer J, Tjonneland A, Overvad K, Jakobsen MU, Boeing H, Buijsse B, Masala G, Palli D, Sorensen TI, Saris WH, Feskens EJ. Dietary fiber and subsequent changes in body weight and waist circumference in European men and women. Am J Clin Nutr. 2010 Feb;91(2):329-36. doi: 10.3945/ajcn.2009.28191. Epub 2009 Dec 16. PMID 20016015
- [Background] Gordon M, Naidoo K, Akobeng AK, Thomas AG. Cochrane Review: Osmotic and stimulant laxatives for the management of childhood constipation (Review). Evid Based Child Health. 2013 Jan;8(1):57-109. doi: 10.1002/ebch.1893. PMID 23878124
- [Background] Lecerf JM, Clerc E, Jaruga A, Wagner A, Respondek F. Postprandial glycaemic and insulinaemic responses in adults after consumption of dairy desserts and pound cakes containing short-chain fructo-oligosaccharides used to replace sugars. J Nutr Sci. 2015 Oct 12;4:e34. doi: 10.1017/jns.2015.22. eCollection 2015. PMID 26495125
- [Background] Liu S, Willett WC, Manson JE, Hu FB, Rosner B, Colditz G. Relation between changes in intakes of dietary fiber and grain products and changes in weight and development of obesity among middle-aged women. Am J Clin Nutr. 2003 Nov;78(5):920-7. doi: 10.1093/ajcn/78.5.920. PMID 14594777
- [Background] Meksawan K, Chaotrakul C, Leeaphorn N, Gonlchanvit S, Eiam-Ong S, Kanjanabuch T. Effects of Fructo-Oligosaccharide Supplementation on Constipation in Elderly Continuous Ambulatory Peritoneal Dialysis Patients. Perit Dial Int. 2016 Jan-Feb;36(1):60-6. doi: 10.3747/pdi.2014.00015. Epub 2014 Oct 7. PMID 25292404
- [Background] Nakamura Y, Nosaka S, Suzuki M, Nagafuchi S, Takahashi T, Yajima T, Takenouchi-Ohkubo N, Iwase T, Moro I. Dietary fructooligosaccharides up-regulate immunoglobulin A response and polymeric immunoglobulin receptor expression in intestines of infant mice. Clin Exp Immunol. 2004 Jul;137(1):52-8. doi: 10.1111/j.1365-2249.2004.02487.x. PMID 15196243
- [Background] Slavin J. Fiber and prebiotics: mechanisms and health benefits. Nutrients. 2013 Apr 22;5(4):1417-35. doi: 10.3390/nu5041417. PMID 23609775
- [Background] van den Heuvel EG, Muijs T, Brouns F, Hendriks HF. Short-chain fructo-oligosaccharides improve magnesium absorption in adolescent girls with a low calcium intake. Nutr Res. 2009 Apr;29(4):229-37. doi: 10.1016/j.nutres.2009.03.005. PMID 19410973
- [Background] van den Heuvel EG, Muys T, van Dokkum W, Schaafsma G. Oligofructose stimulates calcium absorption in adolescents. Am J Clin Nutr. 1999 Mar;69(3):544-8. doi: 10.1093/ajcn/69.3.544. PMID 10075343
- [Background] Vandenplas Y, Zakharova I, Dmitrieva Y. Oligosaccharides in infant formula: more evidence to validate the role of prebiotics. Br J Nutr. 2015 May 14;113(9):1339-44. doi: 10.1017/S0007114515000823. PMID 25989994
- [Background] Ye EQ, Chacko SA, Chou EL, Kugizaki M, Liu S. Greater whole-grain intake is associated with lower risk of type 2 diabetes, cardiovascular disease, and weight gain. J Nutr. 2012 Jul;142(7):1304-13. doi: 10.3945/jn.111.155325. Epub 2012 May 30. PMID 22649266
- [Background] Jenkins AL, Kacinik V, Lyon MR, Wolever TM. Reduction of postprandial glycemia by the novel viscous polysaccharide PGX, in a dose-dependent manner, independent of food form. J Am Coll Nutr. 2010 Apr;29(2):92-8. doi: 10.1080/07315724.2010.10719821. PMID 20679143
- [Background] Wolever TM, Jenkins DJ, Jenkins AL, Josse RG. The glycemic index: methodology and clinical implications. Am J Clin Nutr. 1991 Nov;54(5):846-54. doi: 10.1093/ajcn/54.5.846. PMID 1951155
- [Background] Sheth M, Thakuria A, Chand V and Paban Nath M. Fructooligosaccharide (fos)- a smart strategy to modulate inflammatory marker and lipid profile in non-insulin dependent diabetes mellitus (NIDDM) subjects residing in Assam, India- a randomized control trial. World J Pharma Res, 2015; 4 (5): 2673-2678
- [Background] Yamashita K, Kawai K, Itakura M. Effects of fructo-oligosaccharides on blood glucose and serum lipids in diabetic subjects. Nutr Res, 1984; 4(6):961-6.
- [Derived] Shah P, Wolever TM, Jenkins AL, Ezatagha A, Campbell J, Zurbau A, Jain M, Gote M, Bhaduri A, Mullick A. Acute glycemic and insulin response of Fossence alone, or when substituted or added to a carbohydrate challenge: A three-phase, acute, randomized, cross-over, double blind clinical trial. Heliyon. 2021 Apr 28;7(4):e06805. doi: 10.1016/j.heliyon.2021.e06805. eCollection 2021 Apr. PMID 33997376